CLINICAL TRIAL: NCT03897972
Title: Proof-of-principle Pilot Study to Investigate Whether Online Personalised Dietary Advice Given by the eNutri Diet App Encourages Greater Dietary Behaviour Change Than General Advice in UK Adults After 12 Weeks
Brief Title: Study to Evaluate the 'eNutri' Online Personalised Nutrition App in the United Kingdom (UK)
Acronym: EatWellEUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Director of the Hugh Sinclair Unit of Human Nutrition, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08/19
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Dietary Modification; Dietary Habits
Keywords: Personalised nutrition
MeSH Terms: conditions — Feeding Behavior | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-personalised general diet advice (Active Comparator): Control group to receive non-personalised dietary advice based on general public health dietary recommendations for Northern Europe. Advice will be delivered to the participant via the eNutri web application.
  Interventions: Behavioral: Non-personalised diet advice delivered via the eNutri app (control)
- Personalised diet advice (Experimental): Intervention group to receive personalised dietary advice generated by the eNutri app from their actual dietary intakes and tailored according to their body mass index and food preferences. Advice will be delivered to the participant via the eNutri app web application and will be generated based on their adherence to an 11-item diet quality score suitable for Northern European populations.
  Interventions: Behavioral: Personalised diet advice delivered via the eNutri app (intervention)

INTERVENTIONS:
Behavioral: Non-personalised diet advice delivered via the eNutri app (control) — Non-personalised dietary advice to improve food choices based on standard population guidelines delivered by the eNutri app and irrespective of the dietary intakes from the food frequency questionnaire (control group).
  Arms: Non-personalised general diet advice
Behavioral: Personalised diet advice delivered via the eNutri app (intervention) — Personalised dietary advice to improve food choices based on adherence to an 11-item diet quality score, which is determined by the eNutri app in response to the dietary intakes from the food frequency questionnaire (intervention group).
  Arms: Personalised diet advice

SUMMARY:
The proof-of-principle EatWellEUR pilot study will investigate whether online personalised dietary advice encourages greater dietary behaviour change after 12 weeks compared with general population-based diet advice. Dietary change will be quantified from an 11-item diet quality score (DQS) suitable for Northern European populations that is calculated from the results of the eNutri food frequency questionnaire (FFQ) at baseline and week 12.

DETAILED DESCRIPTION:
The proof-of-principle EatWellEUR pilot study will investigate whether online personalised dietary advice encourages greater dietary behaviour change after 12 weeks compared with general population-based diet advice. Both groups will receive two prompts to remind them of their diet advice at weeks 4 and 8. Dietary change will be quantified from an 11-item diet quality score (DQS) suitable for Northern European populations that is calculated from the results of the eNutri food frequency questionnaire (FFQ) at baseline and week 12. 98 participants will be recruited per study arm and will be randomly allocated to an intervention arm using a minimisation technique integrated with the eNutri app.

ELIGIBILITY:
Inclusion Criteria:

* Living in the UK
* Can understand written English

Exclusion Criteria:

* Food allergies or food intolerances (diagnosed or self-diagnosed)
* Receiving professional nutritional advice from a dietitian, nutritionist or medical professional
* Following a specialised diet (e.g. vegan, calorie-controlled/weight-loss diet)
* Athletes or those following a or sports nutrition regimen
* Pregnant, lactating or planning a pregnancy within the next 3 months
* Diagnosed medical conditions that require specific dietary guidance (e.g. diabetes, Crohn's disease or eating disorders), those who are currently undergoing rigorous medical treatment (e.g. chemotherapy for cancer) or conditions that affect memory (e.g. dementia)
* Medications that impact on diet (e.g. weight-loss medication) or involve dietary restrictions
* Those who eat less than 2 meals per day
* Excessive use of herbal or dietary supplements (e.g. 3 or more per day)
* Taking part in another nutrition study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
eNutri diet quality score (DQS) | Baseline & week 12
  Dietary intake at baseline and week 12 will be assessed via the eNutri food frequency questionnaire (FFQ) from which an 11-item eNutri DQS will be calculated. The eNutri DQS was developed for Northern Europe and quantifies diet quality (i.e. the healthiness of a diet). It is composed of 11 food and nutrient components (contributing 10 points each) that are summed to give an overall score (between 0-110 points), where higher scores reflect the healthiest diets based on adherence to dietary recommendations.

SECONDARY OUTCOMES:
Body mass index (BMI) | Baseline & week 12
  Self reported measurements of weight and height will be used to determine BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lovegrove, Professor, Principal Investigator — Hugh Sinclair Unit of Human Nutrition
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No